CLINICAL TRIAL: NCT00575198
Title: Non-inferiority Randomized Trial Evaluating Removal of Thoracostomy Tubes Independent of the Drainage Amount Versus Removal When the Drainage Amount Is Low
Brief Title: Drainage Amount for Removal of Thoracostomy Tube
Acronym: DARTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200715709
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Pneumothorax; Pleural Effusion
Keywords: Chest tubes; Trauma
MeSH Terms: conditions — Pneumothorax; Pleural Effusion; Wounds and Injuries | interventions — Drainage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): No drainage threshold
  Interventions: Other: No drainage threshold
- 2 (Active Comparator): Drainage <2 mL/kg
  Interventions: Other: Drainage <2 mL/kg

INTERVENTIONS:
Other: No drainage threshold — Removal of the thoracostomy tube independently of the amount of fluid that drained from the tube in the prior 24 hours
  Arms: 1
Other: Drainage <2 mL/kg — Removal of the thoracostomy tube only if the drainage from the tube in the prior 24 hours is less than 2 mL/kg of the patient's ideal body weight
  Other Names: Standard thoracostomy tube management
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether chest tubes can be safely removed without considering how much fluid is draining through the tube.

DETAILED DESCRIPTION:
Thoracostomy tubes are routinely used to drain the pleural space of fluid and gas to optimize pulmonary mechanics. Clinicians frequently postpone removal of thoracostomy tubes if the drainage from the tube exceeds a specific volume threshold for the prior 24 hours. However, there is substantial variability in the drainage volume threshold that different clinicians use, and no threshold has been established as clearly superior to any other. Removing tubes independently of the drainage volume may result in a greater risk of pleural effusion or pneumothorax requiring an invasive drainage procedure. However, removing tubes independently of the drainage volume might also expedite recovery by allowing earlier removal of the tube, thus diminishing pain and increasing patient mobility.

Thoracostomy tube management practices, including the drainage volume threshold used, may be dissimilar for different types of disease processes, so this study will be restricted to patients who required a thoracostomy tube for treatment of traumatic injury.

ELIGIBILITY:
Inclusion Criteria:

* Thoracostomy tube in place for <72 hours
* Age at least 14 years
* Hospitalized for traumatic injury or elective operation

Exclusion Criteria:

* Thoracostomy tube already removed from the pleural cavity of interest
* Mediastinal tubes
* Death expected within 48 hours
* Prisoner status
* Severe congestive heart failure
* End-stage liver disease
* End-stage renal disease
* History of or suspected empyema involving the pleural cavity of interest
* History of or anticipated need for pleurodesis of the pleural cavity of interest
* Malignant pleural effusion
* Pregnancy
* Previous participation in this study
* Thoracostomy tube drainage already <2 mL/kg

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2007-12; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Invasive drainage procedure | Within 60 days

SECONDARY OUTCOMES:
Time to thoracostomy tube removal | Within 60 days
Pulmonary symptoms | 60 days
Mortality | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Garth H Utter, MD MSc, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Medical Center, Sacramento, California, United States